CLINICAL TRIAL: NCT06326151
Title: Study for a Randomised Controlled Trial: Effect of an Interdisciplinary Psycho-educational Intervention Programme on Caregivers of Dependent Older Adults
Brief Title: Interdisciplinary Psychoeducational Intervention Programme for Caregivers of Dependent Older Adults
Status: Not yet recruiting | Phase: Not Applicable | Type: Interventional
Sponsor: University of Salamanca (Other)
Responsible Party: Principal Investigator, Prof. Dr. Eduardo J Fernández Rodríguez, Professor, University of Salamanca
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Supportive Care
Other Study IDs: UMAPS-UDATO
Record Dates: First submitted 2024-03-11; First posted 2024-03-22 (Actual); Last update posted 2024-03-22 (Actual); Status verified 2024-03

CONDITIONS: Dependent Older People; Family Caregiver; Interdisciplinary; Intervention; Occupational Therapy; Psychoeducational; Psychology

STUDY DESIGN:
Who Masked: Outcomes Assessor
Masking Description: The work of sequencing, randomisation, recruitment and allocation of the trial sample will be carried out by research staff who are not involved in the assessments or interventions of each group, thus avoiding any potential bias in the trial.
  Participants will also be blinded and will not know which group they have been allocated to and therefore which intervention they will receive. In order to minimise any contamination between groups, the assessment process will be carried out by external research staff who will perform the measurements and who have been previously trained and educated to avoid subjective bias in the process, as they will be unaware of the intervention group to which they have been assigned, thus masking the blinded assessment by third parties in the clinical trial. In addition, the researchers responsible for the statistical analysis of the trial will be blinded in order to increase the rigour of the trial process and thus the scientific quality.
Oversight: Data Monitoring Committee: Yes | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Health Education Programme (Active Comparator): Why: Upon discharge from the hospital, at the end of the baseline assessment, caregivers will receive instructions and recommendations for maintaining an active and healthy lifestyle. This will be done by encouraging self-care and good practices in caring for their dependent family member, as part of a health education programme. The benefits of an active lifestyle and general guidelines are emphasized.
  What (materials): Instructions and recommendations for a health education programme.
  What (procedures): Participants will receive instructions and recommendations on how to maintain an active and healthy lifestyle, promoting self-care and good practices in caring for their dependent family member.
  How: The caregiver will receive the material individually at the time of referral, before being discharged from the hospital.
  When and for how long: The intervention consists of a single session and details of the time and duration will be provided to participants.
  Interventions: Behavioral: Health Education Programme
- Interdisciplinary Psychoeducational Programme (Experimental): Why: The programme is based on an interdisciplinary psychoeducational intervention from the fields of occupational therapy and psychology.
  What (materials): projector, computer, screen, presentation of content, stationery, chairs, tables and self-recording of home tasks.
  What (procedures): Patients assigned to the experimental group will follow an interdisciplinary psychoeducational programme structured and supervised at the University of Salamanca, consisting of a health education programme combined with an interdisciplinary psychoeducational programme from the perspective of psychology and occupational therapy.
  Who will carry out the interventions: modules: (I) understanding the syndrome or disease and managing difficult everyday caring situations or behaviours, (II) emotions and misconceptions about caring, and (III) self-care (Table 1).
  When and for how long: Each participant will receive 4 sessions per month for 3 months, for a total of 12 sessions.
  Interventions: Behavioral: Interdisciplinary Psychoeducational Programme

INTERVENTIONS:
Behavioral: Interdisciplinary Psychoeducational Programme — This intervention is based on the principle of complementing and integrating both disciplines in order to meet the psychological needs of family carers and to train them in knowledge and strategies aimed at the correct performance of activities of daily living in order to promote the maximum autonomy and functionality of dependent people with cognitive impairment, and that this favours discharge, self-care, improvement of the affective state and quality of life of family carers.
  Arms: Interdisciplinary Psychoeducational Programme
Behavioral: Health Education Programme — Upon discharge from the hospital, at the end of the baseline assessment, caregivers will receive instructions and recommendations for maintaining an active and healthy lifestyle. This will be done by encouraging self-care and good practices in caring for their dependent family member, as part of a health education programme. The benefits of an active lifestyle and general guidelines are emphasized.
  Arms: Health Education Programme

SUMMARY:
Background: Caring for an older dependent adult with cognitive impairment can have negative consequences for the family caregiver. Interdisciplinary interventions are necessary to address their needs jointly and comprehensively. While attempts have been made to improve their situation from different disciplines in isolation, a collaborative approach is required to ensure the best possible outcome.

Methods: A parallel, randomized, controlled clinical trial with two arms will be conducted at the Occupational Therapy Teaching and Care Unit (UDATO) and the Municipal Psychosocial Support Unit for the Elderly (UMAPS), both of which belong to the University of Salamanca and are in agreement with the City Council of Salamanca, Spain. The trial will also be conducted at the University Care Centre of Salamanca (CAUSA). People aged 60 years or older will be recruited as family caregivers of dependent older adults with cognitive impairment in a chronic situation. Participants will be divided into two groups: the intervention group (IG) will carry out an interdisciplinary psychoeducational programme from the perspective of psychology and occupational therapy, and the control group (CG) will carry out a controlled follow-up. Participants will complete 12 sessions over a period of 3 months, followed by three monthly reinforcement sessions after the intervention. At the beginning and end of the intervention, participants will be assessed and socio-demographic data will be collected along with the following scales: the Spanish version of the Caregiver Burden Interview (CBI), the Spanish version of the Center for Epidemiologic Studies-Depression Scale (CES-D), the Psychosocial Support Questionnaire adaptation (PSQ), the General Health Questionnaire (GHQ), the World Health Organization Quality of Life Assessment - AGE (WHOQOL-AGE) and the Bayer-Activities of Daily Living Scale (B-ADL).

Discussion: The objective of this study is to enhance conventional clinical practice for family caregivers of dependent older adults. This will be achieved through an interdisciplinary psychoeducational intervention that aims to reduce overload and depressive symptomatology, increase social support, improve health and perceived quality of life, and enhance understanding of the syndrome/illness. The intervention will also focus on managing difficult situations associated with day-to-day caregiving, managing emotions and associated erroneous beliefs, and promoting self-care. Additionally, the study aims to improve the functionality of the cared-for person.

ELIGIBILITY:
Inclusion Criteria:

* Be the primary family caregiver of a person with cognitive impairment (Mini Mental State Examination (MMSE) < 24 points in a situation of moderate or severe dependency (Barthel) ≤ 55
* Be aged 60 years or older; have been the primary family caregiver for one year or more
* Voluntarily sign the consent form to participate and complete the initial assessment.

Exclusion Criteria:

* Lack of literacy or significant deficits in language comprehension and being a formal carer -
* Receiving financial remuneration for caring for the sick person.

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Enrollment: 70 (Estimated)
Dates: Start 2024-09-01 (Estimated); Primary Completion 2025-09-01 (Estimated); Study Completion 2025-12-31 (Estimated)

PRIMARY OUTCOMES:
Mini Mental State Examination (MMSE) | Baseline; "3 months follow up"; "up to 24 weeks"
  temporal and spatial orientation, fixation, attention and arithmetic, memory, nomination, repetition, comprehension, reading, writing and drawing.
Barthel Index | Baseline; "3 months follow up"; "up to 24 weeks"
  degree of dependency in activities of daily living
Caregiver Burden Interview | Baseline; "3 months follow up"; "up to 24 weeks"
  perceived overload

SECONDARY OUTCOMES:
Centre for Epidemiological Studies Depression Scale | Baseline; "3 months follow up"; "up to 24 weeks"
  depressive symptoms
Adaptation of the Psychosocial Support Questionnaire | Baseline; "3 months follow up"; "up to 24 weeks"
  perceived psychosocial support
General Health Questionnaire | Baseline; "3 months follow up"; "up to 24 weeks"
  perceived health
World Health Organization Assessment of Quality of Life - AGE (WHOQOL-AGE) | Baseline; "3 months follow up"; "up to 24 weeks"
  Quality of Life
The Bayer-Activities of Daily Living Scale (B-ADL) | Baseline; "3 months follow up"; "up to 24 weeks"
  functional disabilities in elderly patients with mild to moderate dementia or cognitive impairment

CONTACTS AND LOCATIONS:
Locations (1):
- Eduardo Jose Fernandez Rodriguez, Salamanca, Castille and León, Spain

IPD SHARING:
Plan to Share IPD: Yes
They will be made available to researchers in the document repository "GREDOS" of the University of Salamanca, Spain.
Supporting Information: Study Protocol, ICF
Time Frame: Data will be available at the end of the study.
Access Criteria: Open access for researchers.
URL: http://gredos.usal.es/

REFERENCES:
- [Derived] Garcia-Tizon SJ, Gomez CS, Martinez MBB, Prados ABN, Rodriguez EJF. Study protocol for a randomised controlled trial: effect of an interdisciplinary psycho-educational intervention programme on caregivers of dependent older adults. BMC Geriatr. 2025 Aug 30;25(1):674. doi: 10.1186/s12877-025-06305-w. PMID 40885892